CLINICAL TRIAL: NCT05506891
Title: Efficacy and Safety of Astragalus for Non-Motor Symptoms of α-Synucleinopathy：an Open-Label Self-Controlled Before-and-After Study
Brief Title: Efficacy and Safety of Astragalus for Non-motor Symptoms of α-Synucleinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS-PDS
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Parkinsonism
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astragalus group (Experimental)
  Interventions: Drug: Astragalus
- Physical therapy group (Active Comparator)
  Interventions: Behavioral: Physical therapy group

INTERVENTIONS:
Behavioral: Physical therapy group — Limit water and sodium intake. Raise the head of the bed. Standardized amount of exercise. Low temperature diet and small meals. Avoid alcohol, coffee and dehydration. The treatment lasted for 3 months.
  Arms: Physical therapy group
Drug: Astragalus — After a 2-week washout period, astragalus granules 15g, drunk with warm water, once a day, will be taken for 3 months.
  Arms: Astragalus group

SUMMARY:
α-Synucleinopathy is a cluster of neurodegenerative disease with motor and non-motor symptom. However, there is still a lack of research on the treatment for non-motor symptoms of α-synucleinopathy, especially autonomic dysfunctions such as orthostatic hypotension. Efficacy and safety of astragalus for non-motor symptoms of α-synucleinopathy will be assessed by an open-label self-controlled before-and-after study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a clinical diagnosis of PD, MSA and DLB, with orthostatic hypotension.
* Participants with cognitive disorder.
* Adults signed informed consents.

Exclusion Criteria:

* Patients with history of astragalus allergy.
* Patients with secondary Parkinsonism that cannot be excluded.
* Patients with diseases that may cause other types of hypotension or similar symptoms/signs because of hypotension
* Patients with other medical conditions requiring treatments that may affect blood pressure.
* Patients with other neurological disorders.
* Patients with serious comorbidities and immune diseases.
* Uncooperative patients.
* Pregnant or lactating women.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline mean arterial pressure after 3 minutes of upright posture versus decubitus position (mmHg) at 3 months. | Baseline vs 3 months after treatment.
  Mean arterial pressure was calculated as ⅓ pulse pressure + diastolic pressure.

SECONDARY OUTCOMES:
OH Questionnaire score | Baseline vs 3 months after treatment.
  ΔHR/ΔSBP means heart rate (HR) and systolic blood pressure (SBP) from baseline OH Questionnaire score
Change from baseline Rate of change in ΔHR/ΔSBP at 3months. | Baseline vs 3 months after treatment.
  ΔHR/ΔSBP means heart rate (HR) and systolic blood pressure (SBP) from baseline lying position to standing for 3 minutes
Change from baseline HRV (ms) at 3months. | Baseline vs 3 months after treatment.
  Heart rate variability (HRV) was calculated as the maximum bpm - minimum bpm.
Change from baseline decumbent and orthostatic digit span (DDS) difference at 3months. | Baseline vs 3 months after treatment.
  DDS is an executive function measurement tool
Change from baseline decumbent and orthostatic character conversion (CDS) difference at 3months. | Baseline vs 3 months after treatment.
  CDS is an executive function measurement tool
Change from baseline MoCA scores at 3 months. | Baseline vs 3 months after treatment.
  The Montreal Cognitive Assessment (MoCA)
Change from baseline CDR scores at 3 months. | Baseline vs 3 months after treatment.
  The Clinical Dementia Rating (CDR)
Change from baseline RAVLT scores at 3 months. | Baseline vs 3 months after treatment.
  The Rey Auditory Verbal Learning Test (RAVLT)
Change from baseline HAS scores at 3 months. | Baseline vs 3 months after treatment.
  The Hamilton Anxiety Scale (HAS)
Change from baseline HDS scores at 3 months. | Baseline vs 3 months after treatment.
  The Hamilton Depression Scale (HDS)
Change from baseline NPI scores at 3 months. | Baseline vs 3 months after treatment.
  The Neuropsychiatric Inventory (NPI)
Change from the baseline plasma α-synuclein levels (ng/ml) at 3 months. | Baseline vs 3 months after treatment.
Change from baseline Vic at 3 months. | Baseline vs 3 months after treatment.
  The intra-cellular compartment (Vic) of the Neurite Orientation Dispersion and Density Imaging (NODDI) model represents diffusion within the axons and cells.
Change from baseline ODI at 3 months. | Baseline vs 3 months after treatment.
  NODDI models the dispersion of axonal fibers with the use of an Orientation Dispersion Index (ODI).
Change from baseline PAF (Hz) at 3 months. | Baseline vs 3 months after treatment.
  The alpha-peak frequency (PAF) is the frequency with the highest power within the alpha-band.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No